CLINICAL TRIAL: NCT04397393
Title: Does Camel Milk Consumption Decrease The Efficacy Of Midazolam For Sedation: A Pilot Study
Brief Title: Does Camel Milk Consumption Decrease The Efficacy Of Midazolam For Sedation
Status: Terminated | Type: Observational
Why Stopped: insufficient data
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Nils Engelmann, Anesthesia Consultant, ART Fertility Clinics LLC
Other Study IDs: 1910-ABU-090-NE
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia; IVF
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-camel milk consumption: non-camel milk consumption over life time
  Interventions: Drug: Midazolam
- camel milk consumption: camel milk consumption at least once during lifetime, with 2 subgroups of camel milk consumption: once, twice, three times; as well as regularly (daily, once per week, once per month, once per year).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Dosage of Midazolam (in mg) needed to achieve satisfactory level of sedation to perform OPU

SUMMARY:
The primary aim is to verify if camel milk consumption has an impact on the amount of Midazolam needed to achieve a satisfactory level of sedation for oocyte retrieval, compared to patients never having consumed camel milk.

DETAILED DESCRIPTION:
A pilot study will be performed on patients undergoing oocyte retrieval (OPU) for the first time, and correlated to camel milk consumption versus never consumed camel milk, as well as age, BMI (body mass index), number of follicles at the time of OPU, number of previous OPUs in other clinics, previous vaginal delivery, past medical history positive for chemo therapy, alcohol consumption, use of prescribed or illicit drugs, or chronic pain medication.

The main objective is to analyse if the consumption of camel milk, the frequency, or lack thereof correlates with the amount of the sedative drug Midazolam needed to achieve an acceptable level of sedation in order to estimate the dosage needed in both patient groups more adequately, reducing either discomfort felt at a too low an initial dosage, as well as avoiding a deeper level of sedation than needed with subsequent prolonged stay in recovery and unpleasant feelings of dizziness and drowsiness, potentially requiring antagonizing Midazolam by the use of Flumazenil, and reducing overall costs and length of stay in recovery and bed occupancy and enhancing patient experience and satisfaction.

Would this study enable the Investigators to determine further effect of camel milk on other drugs used for various other purposes, and lead to a change in dose regimen?

ELIGIBILITY:
Inclusion Criteria:

* Arab origin
* Female 18 -48 years of age
* BMI < 37 kg/m2
* All ovarian stimulation protocols

Exclusion Criteria:

* Previous oocyte retrieval at our center
* Post chemo therapy
* Illicit drug use
* Chronic pain medication
* Medication which is known to increase the activity of liver enzymes
* Any alcohol consumption
* Previous vaginal delivery

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: population is defined by all females of Arab origin, booked for oocyte retrieval for the first time in our center
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Dosage of Midazolam (in mg) needed to achieve satisfactory level of sedation to perform the OPU | 1 day
  Mean dosage of Midazolam for both groups (Camel milk consumption vs no camel milk consumption

CONTACTS AND LOCATIONS:
Overall Officials: Nils Engelmann, MD, Principal Investigator — IVI Middle East Fertility Clinic LLC
Locations (1):
- IVI Middle East Fertility Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Consumption of Camel Milk — http://www.fao.org/3/X6528E/X6528E03.htm#chIII.
- See also: Gast, M., Mauboisj, L. and Adda, J. Le lait et les produits laitiers en Ahaggar. Centr. Rech. Anthr. Prehist. Ethn. 1969 — http://www.fao.org/3/X6528E/X6528E11.htm
- See also: Kuchabaev, K.A. Cherepanova, V.P. and Panomarev P.P. Feeding, milk productivity and chemical composition of camel milk. : 58-62, 1972.El-Bahay, 1962 — http://www.fao.org/3/X6528E/X6528E11.htm
- See also: Kon, S.K. Milk and milk products for human nutrition. FAO Nutrition Serv. 7, p. 6, 1959 (Revised in 1972)., Knoess, K.H. Milk production of the dromedary. In: Camels. IFS Symposium, Sudan. 201-214, 1979 — http://www.fao.org/3/X6528E/X6528E11.htm
- See also: Dhingra, D.R. The component fatty acid and glycerides of the milk fats of Indian goats and sheep. Biochem. J. 27: 851-859, 1933 — http://www.fao.org/3/X6528E/X6528E11.htm
- See also: Dhingra, D.R. Fatty acids and glycerides of the milk fat of camels. Biochem. J. 28: 73-78, 1934 — http://www.fao.org/3/X6528E/X6528E11.htm
- See also: Ohris, S.P. and Joshi, B.K. Composition of camel milk. Indian Vet. J. 38(a): 514-516, 1961; 38(b): 604-606, 1961 — http://www.fao.org/3/X6528E/X6528E11.htm
- See also: Epstein, H. The origin of the domestic animals of Africa. Vol. 2. New York. Africiana Publ. Corp. Leipzig. Edition Leipzig. 1971 — http://www.fao.org/3/X6528E/X6528E11.htm